CLINICAL TRIAL: NCT04377880
Title: Development of Cellular Models for Osteoblast Response Study to Adipocytic Secretions in an Osteoporosis Context.
Acronym: ROSA
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Collaborators: Universite du Littoral Cote d'Opale (Other)
Responsible Party: Sponsor
Other Study IDs: 2019_18R; 2020-A00027-32 (Other: ID-RCB number,ANSM)
Record Dates: First submitted 2020-05-05; First posted 2020-05-06 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Osteoporosis
Keywords: Bone; Osteoporosis; Osteoblast; Adipocyte; Cellular models
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Bone fragments; RNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The recent studies suggest that secretions from medullary adipocytes are involved in the mechanisms of bone loss in osteoporosis (OP) through their actions on neighbouring osteoforming cells, the osteoblasts. The objective of the research is the development of new cellular models representing the aging skeleton to confirm this hypothesis. To this end, osteoblasts will be isolated from human bone fragments coming from femoral heads discarded during total hip replacement surgery. The osteoblastic response to secreted factors released from medullary adipocytes of commercial origin will be analysed using conditioned media incubations. This phenotypic response will be quantified for each subject through the analysis of gene expression levels. Inter-subject phenotype variations will be related to bone density and microarchitecture data obtained by X-ray microtomography. This will assess the existence of a correlation between the osteoblast response to adipocyte secretions and the degree of osteoporosis of the subject from whom the cells are derived.

ELIGIBILITY:
Inclusion Criteria:

* Adult subject
* Surgical indication for hip prosthesis implantation
* Affiliation to a social insurance regime

Exclusion Criteria:

* Rejection of participation
* Diagnosed bone diseases other than osteoarthritis or osteoporosis
* Cancer
* Pregnant Women
* Subject under guardianship or trusteeship
* Subject unable to understand the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a surgical indication for a prosthetic hip joint at the Boulogne-sur-Mer hospital.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2024-09-04 (Actual); Study Completion 2024-09-04 (Actual)

PRIMARY OUTCOMES:
the level of gene expression of adipocyte markers such as PPARG and leptin | Baseline
  The effect of adipocyte secretion products on osteoblasts will be evaluated by incubating osteoblasts from human bone biopsies with commercially available adipocyte conditioned cell media. Phenotypic changes in osteoblastic cells will then be evaluated by analyzing their gene expression profile and comparing them with those of osteoblasts incubated in unconditioned media. The selected criteria for judging osteoblast alteration will be the measurement of the level of gene expression of adipocyte markers such as PPARG and leptin.

SECONDARY OUTCOMES:
Inter-subject phenotype variations by X-ray microtomography | Baseline
  Inter-subject phenotype variations will be related to quantitative bone microarchitecture data determined by X-ray microtomography.

CONTACTS AND LOCATIONS:
Overall Officials: Eric FODZO, MD, Principal Investigator — University Hospital, Lille
Locations (1):
- Centre hospitalier, Boulogne-sur-Mer, France